CLINICAL TRIAL: NCT06482359
Title: A Phase 3, Randomized, Observer-Blinded, Study to Compare the Safety and Immunogenicity of 3 Lots of SARS-CoV-2 rS Nanoparticle and Trivalent Hemagglutinin Nanoparticle Influenza Combination Vaccine With Matrix M™ Adjuvant in Participants ≥ 65 Years of Age
Brief Title: Lot Consistency Study of COVID-19 and Influenza Combination Vaccine
Acronym: CIC
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: It was decided to not move forward with the study.
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CIC-E-303
Record Dates: First submitted 2024-06-27; First posted 2024-07-01 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Influenza
Keywords: COVID-19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lot 1 (Group 1) (Active Comparator): CIC vaccine will be administered as a single 0.5 mL IM injection in the deltoid on Day 0
  Interventions: Biological: coformulated CIC Vaccine
- Lot 2 (Group 2) (Active Comparator): CIC vaccine will be administered as a single 0.5 mL IM injection in the deltoid on Day 0
  Interventions: Biological: coformulated CIC Vaccine
- Lot 3 (Group 3) (Active Comparator): CIC vaccine will be administered as a single 0.5 mL IM injection in the deltoid on Day 0
  Interventions: Biological: coformulated CIC Vaccine
- Fluzone HD (Active Comparator): Fluzone HD trivalent will be administered as a suspension 1M Injection at 0.5mL on Day 0
  Interventions: Biological: Fluzone HD trivalent

INTERVENTIONS:
Biological: coformulated CIC Vaccine — SARS-CoV-2 rS (35 µg) + trivalent hemagglutinin nanoparticle influenza (tNIV) antigen (180 µg; 60 µg per strain) + Matrix-M adjuvant (75 µg)
  Other Names: SARS-CoV-2 rS, tNIV, Matrix-M adjuvant
  Arms: Lot 1 (Group 1); Lot 2 (Group 2); Lot 3 (Group 3)
Biological: Fluzone HD trivalent — 60 µg per strain of 3 strains (sodium phosphate buffered isotonic sodium chloride solution + formaldehyde and octyl phenol ethoxylate)
  Arms: Fluzone HD

SUMMARY:
The goal of Phase 3 Study is Comparing the Safety and Immune Response of Three Batches of a COVID-19 and Flu Combination Vaccine in Seniors Aged 65+

DETAILED DESCRIPTION:
This is a randomized, Phase 3 study comparing the safety and immunogenicity of 3 different lots of Novavax coronavirus disease 2019 (COVID-19) and influenza combination (CIC) vaccine in terms of wild-type influenza hemagglutinin inhibition (HAI) antibody responses to 3 vaccine-homologous influenza strains (i.e., 2 influenza A strains and an influenza B-Victoria lineage strain) and 1 IM dose of Fluzone HD in terms of the neutralizing antibody (NAb) responses to the homologous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) strain.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all the following criteria:

1. Willing and able to give informed consent prior to study enrollment.
2. Medically stable adult male or female ≥ 60 years of age at Screening.
3. Participants may have 1 or more chronic medical diagnoses, but should be clinically stable as assessed by:

   1. Absence of changes in medical therapy in the past 2 months due to treatment failure or toxicity.
   2. Absence of medical events qualifying as SAEs within 3 months; and
   3. Absence of known, current, and life-limiting diagnoses which render survival to completion of the protocol unlikely in the opinion of the Investigator.
4. The participant has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at Screening.
5. Participant must be able to receive an injection in the deltoid of either arm.
6. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AEs.
7. Participants must have completed a primary vaccination series/booster against SARS-CoV-2 with an authorized/approved COVID-19 vaccine, with receipt of last dose of authorized/approved vaccine (with or without boosters[s]) ≥ 8 weeks prior to vaccination.
8. Participants must agree to not participate in any other SARS-CoV-2 or influenza prevention or treatment studies for the duration of the study.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. History of laboratory-confirmed (by polymerase chain reaction [PCR] or rapid antigen test) COVID-19 or asymptomatic SARS-CoV-2 infection; either occurring ≤ 8 weeks prior to Screening.
2. Any ongoing, symptomatic acute illness requiring medical or surgical care or chronic illness that required substantive changes in medication in the past 2 months prior to Screening indicating that chronic illness/disease is not stable (at the discretion of the Investigator). This includes any current workup of undiagnosed illness that could lead to a new condition.
3. Serious chronic diseases inclusive of:

   1. Uncontrolled hypertension;
   2. Congestive heart failure requiring hospitalization within 3 months prior to Screening;
   3. Chronic obstructive pulmonary disease (COPD) requiring hospitalization within 3 months prior to Screening;
   4. Within 3 months prior to Screening, evidence of unstable coronary artery disease as manifested by cardiac interventions (e.g., cardiac stent placement, coronary artery bypass graft surgery), new cardiac medications for control of symptoms, or unstable angina.
   5. Hospitalization for diabetic ketoacidosis within 6 months prior to Screening
   6. Chronic kidney disease/renal requiring institution of substantive new therapy within 3 months prior to Screening
   7. Chronic clinically significant gastrointestinal and hepatic diseases requiring hospitalization or institution of substantive new therapy within 3 months prior to Screening.
   8. Chronic neurological diseases or neurological compromise preventing access to the study clinic, compliance with protocol, or accurate reporting of safety.
4. Participation in research involving an investigational product (drug/biologic/device) within 90 days before planned date of vaccination.
5. Use of COVID-19 prophylactic or treatment monoclonal antibodies or antibody cocktails within 90 days prior to planned date of vaccination.
6. History of a serious reaction to a prior influenza vaccination or known allergy to constituents of influenza vaccines - including egg proteins - or polysorbate 80; or any known allergies to products contained in the investigational product.
7. Any history of anaphylaxis to any prior vaccine.
8. History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine.
9. Receipt of any vaccine in the 4 weeks preceding the study vaccination and any influenza vaccine within 2 months preceding the study vaccination. Note: Routine vaccinations will not be allowed until after study Day 28 and COVID-19 and influenza vaccination will not be allowed until after Day 28.
10. Any known or suspected autoimmune or immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
11. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccines. An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted.
12. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
13. Active cancer (malignancy) therapy within 1 year prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo malign and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the Investigator).
14. Women of childbearing potential (defined as any female participant who is NOT surgically sterile [i.e., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months].
15. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to study vaccination, which in the opinion of the Investigator, might interfere with protocol compliance.
16. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥ 38.0°C, on the planned day of vaccine administration).
17. History of myocarditis or pericarditis.
18. Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
19. Study team member or immediate family member of any study team member (inclusive of Sponsor, contract research organization [CRO], and study site personnel involved in the conduct or planning of the study).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-11-16 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with solicited local and systemic AEs. | 7 days post-vaccination]
  Numbers of participants with solicited local and systemic AEs over the 7 days post-vaccination.
Numbers of participants reporting Unsolicited AEs and medically attended adverse events (MAAEs). | 28 days post-vaccination.
  Numbers of participants reporting unsolicited AEs and medically attended adverse events (MAAEs) over 28 days post-vaccination.
Number of participants with MAAEs, SAEs, AESIs (including [PIMMCs] and myocarditis and/or pericarditis). | 6 months (approximately 182 days) post-vaccination.
  Numbers of participants with Medical Attended Adverse Events (MAAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) (including potential immune-mediated medical conditions [PIMMCs] and myocarditis and/or pericarditis).

SECONDARY OUTCOMES:
Hemagglutination-inhibition (HAI) antibody titers specific for the Hemagglutinin (HA) receptor binding domains of vaccine homologous Influenza A and B strains expressed as Geometric Mean Titer (GMT) | Day 0 to Day 28
  HAI antibody titers specific for the Hemagglutinin (HA) receptor binding domains of vaccine response to immunization of 3 lots of CIC vaccine to 3 vaccine-homologous influenza strains at Days 0 and 28 Expressed as GMT
HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A and B strains expressed as Geometric Mean Fold Rise (GMFR) | Day 0 to Day 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response to immunization of 3 lots of CIC vaccine to 3 vaccine-homologous influenza strains at Days 0 and 28 Expressed as GMFR.
HAI antibody titers specific for the HA receptor binding domains of vaccine homologous Influenza A and B strains expressed as Geometric Mean Titer Ratio (GMTR) | Day 0 to Day 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response to immunization of 3 lots of CIC vaccine to 3 vaccine-homologous influenza strains at Days 0 and 28 Expressed as GMTR
HAI antibody Titers specific for the Hemagglutinin (HA) receptor binding domains of vaccine- homologous influenza strains A and B Expressed as Seroconversion Rate (SCR) | Day 0 to Day 28
  HAI antibody titers specific for the HA receptor binding domains of vaccine response to immunization of 3 lots of CIC vaccine to 3 vaccine-homologous influenza strains at Days 0 and 28 Expressed as SCR.
Neutralizing Antibody (NAb)specific to vaccine homologous wild-type influenza strains A and B Expressed as GMT. | Day- 0 to 28
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay CIC vaccine Expressed as GMT
Neutralizing Antibody (NAb)specific to vaccine homologous wild-type influenza strains A and B Expressed as GMFR. | Day- 0 to 28
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay CIC vaccine Expressed as GMFR.
Number of participants of Neutralizing antibody titers specific to vaccine-matched wild-type A and B influenza strains expressed as GMTR. | Day- 0 to 28
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay CIC vaccine Expressed as GMTR
Percentage of Participants with a Neutralizing Antibody (NAb)specific to vaccine homologous wild-type influenza strains A and B expressed as SCR. | Day- 0 to 28
  Neutralizing antibody titers specific to vaccine homologous wild-type A and B influenza strains, as measured by a neutralization assay CIC vaccine Expressed as SCR